CLINICAL TRIAL: NCT02922166
Title: Effects of SRX246, a Vasopressin Receptor (V1a) Antagonist, on an Experimental Model of Fear and Anxiety in Humans
Brief Title: Effects of SRX246 on an Experimental Model of Fear and Anxiety in Humans
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azevan Pharmaceuticals (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVN012; T-M-1970 (Other: National Institute of Mental Health); NCT03036397 (obsolete NCT alias)
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Fear; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — SRX246

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SRX246 (Experimental): SRX246 oral dosage capsules, daily dose to be taken bid, for up to 7 days
  Interventions: Drug: SRX246
- Placebo (Placebo Comparator): Placebo oral dosage capsules, daily dose to be taken bid, for up to 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRX246 — oral capsule
  Arms: SRX246
Drug: Placebo — oral capsule
  Arms: Placebo

SUMMARY:
To determine the effects of SRX246 on fear and anxiety based on fear-potentiated startle in humans. Additionally, the effects of the compound on emotion recognition will be explored.

DETAILED DESCRIPTION:
The study will use a double-blind, cross-over design in which each subject will receive placebo and SRX246 for 5-7 days before testing (given in counter-balanced order). The study will examine the effect of the drug on the potentiation of startle using a well-established paradigm that involves anticipation of no-shock, predictable shock, and unpredictable shock. Drug effects on emotion recognition will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, ages 21-50, inclusive.
* Subjects able to give their consent and have signed informed consent forms indicating that they understand the purpose and procedures of the study and are willing to participate in the study procedures and restrictions.
* Body mass index (BMI) of 18.5 to 34.0 kg/m2, inclusive, and a total body weight of >50kg (110 pounds).

Exclusion Criteria:

* Non-English speakers
* Current or history of Axis I psychiatric disorder(s) as identified with the Structured Clinical Interview for DSM-IV-TR, non-patient edition (SCID-np) and clinical evaluation.
* Active or history of active suicidal ideation.
* Lifetime alcohol or drug dependence according to the Structured Clinical Interview for DSM-IV-TR, non-patient edition (SCID-np).
* All prescription and non-prescription medications and herbal remedies are prohibited within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication and until at least 7 days or 5 half-lives (whichever is longer) after last dose of study medication, except hormonal contraceptives in females.
* Clear evidence of a first-degree relative with history of psychosis, bipolar disorder or major depression as determined by the family history method; specifically, participant will know diagnosis or treatment in order to confirm presence of disorder.
* Subject is currently participating in another clinical trial in which (s)he is or will be exposed to an investigational or non-investigational drug or device, or has done so within the preceding month.
* Current evidence or history of significant medical illness or organic brain impairment, including syndrome of inappropriate antidiuretic hormone secretion (SIADH), diabetes insipidus (DI), stroke, epilepsy, CNS tumor, demyelinating disease, cardiac, pulmonary, gastrointestinal, renal or hepatic impairment that would likely interfere with the action, absorption, distribution, metabolism, or excretion of SRX246, or influence psychophysiological responses.
* Current evidence of median nerve entrapment or carpal tunnel syndrome.
* Any laboratory abnormality that in the investigators' judgment is considered to be clinically significant (ECG, TSH, LFT, etc.).
* Abnormal urine specific gravity (below 1.00 or above 1.03) as documented by urine sample refractometry.
* Subject who has resting blood pressure outside of a systolic blood pressure range of 90-140 mmHg or a diastolic blood pressure outside a range of 50-90 mmHg on two consecutive measurements taken up to 10 minutes apart.
* Subject who has resting pulse rate greater than 100 bpm or less than 50 bpm on two consecutive measurements taken up to 10 minutes apart.
* Consumption of illicit substances or positive urine toxicology screen throughout the study.
* Pregnancy, lactating/breastfeeding, or positive pregnancy test.
* A history of significant drug allergy or systemic allergic disease (e.g., urticaria, atopic dermatitis), or any known/suspected hypersensitivity to SRX246, or allergy to gelatin.
* Lack of measurable startle response (3 times the baseline EMG activity) for all 9 startles used during the habituation visit.
* Subjects who would be noncompliant with the visit schedule or study procedures. Possible noncompliance may include planned vacations or planned hospitalizations during the study.
* For women who are able to get pregnant and men who are able to father a child, unwillingness to use at least two effective birth control methods for 15 days prior to the time they enroll in the study, and for 15 days after their last exposure to the study drug. Effective methods of contraception for this study include:

  1. hormonal contraception (birth control pills, injected hormones or vaginal ring),
  2. intrauterine device,
  3. barrier methods (condom or diaphragm) combined with spermicide, and
  4. surgical sterilization (hysterectomy, tubal ligation, or vasectomy).
* Employee of NIMH or an immediate family member who is a NIMH employee

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in startle reflex between SRX246 and Placebo | up to 7 days
  Subjects will be exposed to none (N), predictable (P) and unpredictable (U) acoustic and electric shocks.

SECONDARY OUTCOMES:
Change in emotional expression recognition between SRX246 and Placebo | up to 7 days
  Subjects will be shown pictures of faces exhibiting anger, disgust, fear, happiness, sadness and surprise.
Change in State Anxiety Scale between SRX246 and Placebo | up to 7 days
  Subjects will rate their anxiety level during assessments using a self-administered rating scale.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and samples will be shared with Azevan Pharmaceuticals Inc., its affiliates and research partners working with Azevan Pharmaceuticals Inc.